CLINICAL TRIAL: NCT00005775
Title: Randomized Controlled Trial of Parenteral Glutamine Supplementation for Extremely-Low-Birth-Weight (ELBW) Infants
Brief Title: Glutamine Supplementation to Prevent Death or Infection in Extremely Premature Infants
Acronym: Glutamine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Brenda B. Poindexter, Lead Principal Investigator, Indiana University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0020; U10HD027856 (NIH); U10HD021364 (NIH); U10HD034216 (NIH); U10HD034167 (NIH); U10HD021397 (NIH); U10HD027853 (NIH); U10HD027871 (NIH); U10HD021415 (NIH); U10HD027904 (NIH); U10HD027881 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027880 (NIH); U10HD021373 (NIH); U01HD036790 (NIH); M01RR008084 (NIH); M01RR006022 (NIH); M01RR000750 (NIH); M01RR000997 (NIH); M01RR000070 (NIH); M01RR001032 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Sepsis
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW) infants; Prematurity; Glutamine; Total parenteral nutrition; Nutrition; Very low birth weight (VLBW) infants
MeSH Terms: conditions — Premature Birth; Sepsis; Hyperphagia | interventions — Glutamine; amino-acid, glucose, and electrolyte solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glutamine (Experimental): TrophAmine (B. Braun/McGaw) with cysteine hydrochloride (40mg/gm amino acids) with L-glutamine added (20% of the total amount of amino acids)
  Interventions: Drug: Glutamine
- Placebo (Placebo Comparator): Standard TrophAmine (B. Braun/McGaw) with cysteine hydrochloride (40mg/gm amino acids)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glutamine — Infants randomized to glutamine supplementation will receive glutamine any time that parenteral nutrition is required during the first 120 days of hospitalization.
  Other Names: L-Glutamine; TrophAmine
  Arms: Glutamine
Drug: Placebo — TrophAmine given any time that parenteral nutrition is required during the first 120 days of hospitalization.
  Other Names: TrophAmine
  Arms: Placebo

SUMMARY:
This large multicenter double-masked clinical trial tested whether supplementation of standard neonatal parenteral nutrition with glutamine would reduce the risk of death or late-onset sepsis in extremely-low-birth-weight (ELBW, less than or equal to 1000 gm) infants. Neonates with birth weights of 401-1000gm were randomized to standard TrophAmine or TrophAmine supplemented with glutamine before 72 hours and continued until the infants are tolerating full enteral feedings.

DETAILED DESCRIPTION:
Meeting the protein and energy requirements of extremely premature infants in early postnatal life requires early hyperalimentation and the gradual introduction of enteral feedings. Glutamine, which is the most abundant amino acid in the human body and taken up in greatest quantity by the fetus from the placenta, is not routinely provided in neonatal parenteral nutrition preparations.

This large multicenter double-masked clinical trial tested whether supplementation of standard neonatal parenteral nutrition with glutamine would reduce the risk of death or late-onset sepsis in extremely-low-birth-weight (ELBW, less than or equal to 1000 gm) infants. Neonates with birth weights of 401-1000gm were randomized to standard TrophAmine or TrophAmine supplemented with glutamine before 72 hours and continued until the infants are tolerating full enteral feedings.

Infants received a neurodevelopmental assessment by masked, certified examiners at 18-22 months postmenstrual age.

ELIGIBILITY:
Inclusion Criteria:

* 401-1000 gm
* More than 12 hrs and less than 72 hrs after birth; intravenous access
* Parental consent

Exclusion Criteria:

* One or more major congenital anomalies
* Infants meeting criteria for terminal illness
* Congenital nonbacterial infection with overt signs at birth

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1433 (Actual)
Dates: Start 1999-07; Primary Completion 2000-12 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Death or late-onset sepsis | At hospital discharge

SECONDARY OUTCOMES:
Tolerance of enteral feeding (number of days to reach full enteral feeds) and decrease number of episodes of feeding intolerance | At hospital discharge
Necrotizing Enterocolitis | At hospital discharge
Episodes of late-onset sepsis | At hospital discharge
Growth (days to reach 1500 grams) | At hospital discharge
Number of days on parenteral nutrition | At hospital discharge
Length of stay in NICU | At hospital discharge
Neurodevelopmental outcome | 18-22 months corrrected age
Levels of pro-inflammatory cytokines | In the perinatal period

CONTACTS AND LOCATIONS:
Overall Officials: Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Avroy A. Fanaroff, MD, Principal Investigator — Case Western Reserve University; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Barbara J. Stoll, MD, Principal Investigator — Emory University; Charles R. Bauer, MD, Principal Investigator — University of Miami; Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; W. Kenneth Poole, PhD, Principal Investigator — RTI International; David K. Stevenson, MD, Principal Investigator — Stanford University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Jon E. Tyson, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Abbot R. Laptook, MD, Principal Investigator — University of Texas Southwestern Medical Center; Seetha Shankaran, MD, Principal Investigator — Wayne State University; William Oh, MD, Principal Investigator — Women and Infants Hospital, Brown University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - RTI International, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Result] Poindexter BB, Ehrenkranz RA, Stoll BJ, Koch MA, Wright LL, Oh W, Papile LA, Bauer CR, Carlo WA, Donovan EF, Fanaroff AA, Korones SB, Laptook AR, Shankaran S, Stevenson DK, Tyson JE, Lemons JA; National Institute of Child Health and Human Development Neonatal Research Network. Effect of parenteral glutamine supplementation on plasma amino acid concentrations in extremely low-birth-weight infants. Am J Clin Nutr. 2003 Mar;77(3):737-43. doi: 10.1093/ajcn/77.3.737. PMID 12600870
- [Result] Poindexter BB, Ehrenkranz RA, Stoll BJ, Wright LL, Poole WK, Oh W, Bauer CR, Papile LA, Tyson JE, Carlo WA, Laptook AR, Narendran V, Stevenson DK, Fanaroff AA, Korones SB, Shankaran S, Finer NN, Lemons JA; National Institute of Child Health and Human Development Neonatal Research Network. Parenteral glutamine supplementation does not reduce the risk of mortality or late-onset sepsis in extremely low birth weight infants. Pediatrics. 2004 May;113(5):1209-15. doi: 10.1542/peds.113.5.1209. PMID 15121931
- [Result] Oh W, Poindexter BB, Perritt R, Lemons JA, Bauer CR, Ehrenkranz RA, Stoll BJ, Poole K, Wright LL; Neonatal Research Network. Association between fluid intake and weight loss during the first ten days of life and risk of bronchopulmonary dysplasia in extremely low birth weight infants. J Pediatr. 2005 Dec;147(6):786-90. doi: 10.1016/j.jpeds.2005.06.039. PMID 16356432
- [Result] Poindexter BB, Langer JC, Dusick AM, Ehrenkranz RA; National Institute of Child Health and Human Development Neonatal Research Network. Early provision of parenteral amino acids in extremely low birth weight infants: relation to growth and neurodevelopmental outcome. J Pediatr. 2006 Mar;148(3):300-305. doi: 10.1016/j.jpeds.2005.10.038. PMID 16615955
- [Result] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Wright LL, Langer JC, Poole WK; NICHD Neonatal Research Network. Beneficial effects of breast milk in the neonatal intensive care unit on the developmental outcome of extremely low birth weight infants at 18 months of age. Pediatrics. 2006 Jul;118(1):e115-23. doi: 10.1542/peds.2005-2382. PMID 16818526
- [Result] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Higgins RD, Langer JC, Poole WK; National Institute of Child Health and Human Development National Research Network. Persistent beneficial effects of breast milk ingested in the neonatal intensive care unit on outcomes of extremely low birth weight infants at 30 months of age. Pediatrics. 2007 Oct;120(4):e953-9. doi: 10.1542/peds.2006-3227. PMID 17908750
- [Result] Meinzen-Derr J, Poindexter B, Wrage L, Morrow AL, Stoll B, Donovan EF. Role of human milk in extremely low birth weight infants' risk of necrotizing enterocolitis or death. J Perinatol. 2009 Jan;29(1):57-62. doi: 10.1038/jp.2008.117. Epub 2008 Aug 21. PMID 18716628
- [Result] Peralta-Carcelen M, Moses M, Adams-Chapman I, Gantz M, Vohr BR; NICHD Neonatal Research Network; National Institutes of Health. Stability of neuromotor outcomes at 18 and 30 months of age after extremely low birth weight status. Pediatrics. 2009 May;123(5):e887-95. doi: 10.1542/peds.2008-0135. PMID 19403482
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/
- See also: Click here for the Cochrane review "Glutamine supplementation for preventionof morbidity in the preterm infant." — http://www.ncbi.nlm.nih.gov/pubmed/15674878
- See also: NICHD Pregnancy & Perinatology Branch — https://www.nichd.nih.gov/about/org/der/branches/ppb/Pages/overview.aspx